CLINICAL TRIAL: NCT06720012
Title: Total Knee Arthroplasty Inserted With Patient Specific or Standard Instruments
Brief Title: Does the Use of Patient Specific Instrumentation Improve Outcomes in Knee Arthroplasty Surgery for Osteoarthritis When Compared to Standard Posterior Referenced Instrumentation?
Acronym: PRIPSI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Zimmer Biomet (Industry); Ingabritt och Arne Lundbergs Forskningsstiftelse (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53; 210-13 (Other: Regional Ethics Authority Göteborg)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Primary Osteoarthritis Patients Scheduled for Total Knee Replacement Surgery; Osteoarthritis (OA) of the Knee
Keywords: Patient Specific Instrumentation; Total Knee Arthroplasty; Zimmer PSI; NexGen; Materialise
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patient Specific Instrumentation (PSI) (Experimental): PSI cutting guides modeled from a MRI preoperatively and based on the patients unique anatomy.
  Interventions: Device: Patient specific instrumentation (PSI); Procedure: Cemented Total Knee Arthroplasty
- Conventional Instrumentation (Active Comparator): Conventional jig-based intra- and extramedullary instrumentation for the NexGen Knee System.
  Interventions: Device: Conventional instruments; Procedure: Cemented Total Knee Arthroplasty

INTERVENTIONS:
Device: Patient specific instrumentation (PSI) — Cutting guides that are manufactured using advanced imaging and modelling techniques to create instruments that align more closely with the unique anatomy of each patient. Custom guides were created based on a preoperative MRI protocol (Zimmer Patient Specific Instrumentation for NexGen® Complete Knee Solution, Zimmer Biomet, Warsaw, Indiana, United States in collaboration with Materialise NV, Leuven, Belgium) to optimize the placement of the components without the need for intramedullary alignment.
  Other Names: Patient specific cutting guides; Patient-specific guides; Custom instrumentation; Extramedullary femoral cutting system; Patient-matched instruments
  Arms: Patient Specific Instrumentation (PSI)
Device: Conventional instruments — Instruments specific to the implant that are used to guide bone cutting in reference to the intramedullary canal or using an extramedullary jig.
  Other Names: Traditional jig-based instruments; Traditional cutting guides; Jig-based instrumentation; Intra- and extramedullary cutting guides
  Arms: Conventional Instrumentation
Procedure: Cemented Total Knee Arthroplasty — A cemented TKA (NexGen® Complete Knee Solution, Zimmer Biomet, Warsaw, Indiana, United States) is used in all cases with a cruciate retaining (CR) or posterior stabilized (LPS) prosthesis as determined by the surgeon.

SUMMARY:
The goal of this randomized study is to see if using patient-specific instruments (PSI) during total knee replacement surgery improves outcomes compared to standard instruments. The study focuses on adults with knee osteoarthritis who need knee replacement surgery. Specifically, it aims to answer the following questions:

Does using PSI improve knee function and stability as experienced by the patient? Does PSI lead to more normal knee motion during bending and straightening? Does PSI result in at least as good tibial (shin bone) component fixation as standard instruments? Is PSI more cost-effective than standard instruments? Researchers will compare PSI with standard instruments in 70 patients. Half will receive knee replacement surgery using PSI, and the other half with standard instruments. Patients will be randomly assigned to each group.

Participants will:

Undergo knee replacement surgery with either PSI or standard instruments. Have a series of follow-ups, including assessments of knee function, satisfaction, and alignment of the knee implant, conducted before surgery and at 3 months, 1 year, 2 years, and 5 years after surgery.

The study will include patients aged 40-75 with primary osteoarthritis, a body mass index (BMI) below 35, and no other major medical conditions that could impact surgery. Patients will also need to be willing to undergo necessary imaging, such as magnetic resonance imageing (MRI) scans and standing X-rays.

Outcomes will be measured using various assessment tools, including the Oxford Knee Score, Knee Society Score, and a patient satisfaction survey. Researchers will also record surgery details, such as operating time, blood loss, and knee implant size. Imaging methods, including MRI, computed tomgraphy (CT) scans, and specialized X-rays, will be used to evaluate knee alignment and stability over time.

The results of this study are expected to provide insights into whether patient-specific instruments offer clinical or economic advantages over traditional tools in knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Medial or lateral primary osteoarthritis (OA) Ahlbäck Grade 2-4
* Varus or valgus deformity ≤10 degrees, extension defect ≤10 degrees
* Age 40-75 years
* BMI <35
* American Society of Anesthesiologists (ASA) score 1-3.
* Coming from independent living in own home
* Able and willing to undergo MRI scan (for custom patients), full-leg standing radiographs and follow up with RSA
* Written informed consent.

Exclusion Criteria:

* Cortisone treatment during the last 6 months before operation
* Neurological diseases with symptoms, stroke with sequel
* Endocrine diseases with symptoms
* OA secondary to trauma, infection, inflammatory disease or congenital and acquired deformities
* BMI >=35
* OA of the hip with symptoms
* Ongoing infection
* Any metal within 150 mm from the joint line on the side to become operated
* Unable or unwilling to participate in the follow-up.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | Prior to and 2 years post surgery
  A instrument validated for use in Sweden for measuring patient reported functional outcomes following knee arthroplasty. The OKS is widely used due to its reliability and sensitivity to clinically meaningful improvements in knee function after TKA. The score ranges from 12-48 points with a minimal important change of 8 and a ceiling reported to be around 44-48 points.

SECONDARY OUTCOMES:
Knee Society Knee Score (KSKS) | Prior to and up to 5 years post surgery
  A clinician-rated tool that evaluates knee stability and function in activities of daily living. The KSKS is divided into two parts, Knee and Function, each with a max score of 100 points. The minimal clinically important difference of the KSKS is reported to be around 4-10 points for each individual part and a 39-40 increase is considered a substantial clinical improvement.
Oxford Knee Score (OKS) | Prior to and up to 5 years post surgery
  See primary outcome measure.
EuroQol EQ-5D-3L | Prior to and up to 5 years post surgery
  A generic health status measure that allows for the comparison of TKA outcomes across different populations and facilitates cost-effectiveness analyses based on quality-adjusted life years (QALYs). The instrument contains a set of questions reported on a Likert scale which is then converted to a total between 0 and 1 using a value set. The minimal clinically important difference has been reported at 0.0085.
Pain and Patient Satisfaction Visual Analogue Scales (VAS) | (Prior to) and up to 5 years post surgery
  Provides additional patient-centred measures of perceived pain relief and satisfaction with the procedure. The scores are reported on a 0-5 and 0-100 scale.
Radiographic evaluation | Postoperatively, up to three months postop.
  Conventional imaging in the anteroposterior (AP) and lateral views, along with full-leg standing radiographs and CT-scan. These images will be used to assess postoperative alignment and the positioning of TKA components in three planes-coronal, sagittal, and axial (rotational).
Radiographic evaluation, radiolucent lines | Up to 5 years post surgery
  Areas of decreased density (radiolucency) between the bone and cement interface. These are monitored as a potential indicator of loosening or poor fixation.
Radiostereometric Analysis (RSA) | Up to 5 years post surgery
  Used to quantify implant migration as a surrogate marker for fixation stability. Radiologically measures the migration of tantalum markers inserted in the bone in reference to the metal implants.

OTHER OUTCOMES:
Number of patients undergoing revision surgery | Up to 5 years post surgery
  Will be reported as descriptive elements.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no formal IPD plan but we are open to sharing data upon formal request.

REFERENCES:
- [Background] Nunley RM, Ellison BS, Zhu J, Ruh EL, Howell SM, Barrack RL. Do patient-specific guides improve coronal alignment in total knee arthroplasty? Clin Orthop Relat Res. 2012 Mar;470(3):895-902. doi: 10.1007/s11999-011-2222-2. Epub 2011 Dec 20. PMID 22183477
- [Background] Ast MP, Nam D, Haas SB. Patient-specific instrumentation for total knee arthroplasty: a review. Orthop Clin North Am. 2012 Nov;43(5):e17-22. doi: 10.1016/j.ocl.2012.07.004. Epub 2012 Sep 10. PMID 23102417